CLINICAL TRIAL: NCT06037382
Title: Using a Smartphone App to Target Current Mental Health Symptoms of Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: Norris Cotton Cancer Center (Other)
Responsible Party: Principal Investigator, Nicholas Jacobson, Assistant Professor of Biomedical Data Science and Psychiatry, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00032649
Record Dates: First submitted 2023-07-31; First posted 2023-09-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Depression; Anxiety; Cancer
Keywords: Cancer Prevention; Passive sensing
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MoodTriggers App (Experimental): Mood Triggers provides personalized feedback on individuals' maintenance factors (i.e., "triggers") of their anxiety and depressive symptoms based on the theory that such feedback will lead to symptom reduction. Mood Triggers delivers ultra-brief interventions (less than 2 minutes long) where participants view videos which introduce an important skill to treat their anxiety and depressive.
  Interventions: Other: Mood Triggers App

INTERVENTIONS:
Other: Mood Triggers App — The current intervention will deploy a smartphone application called Mood Triggers. Mood Triggers was designed to provide personalized feedback on individuals' maintenance factors (i.e., "triggers") of their anxiety and depressive symptoms based on the theory that such feedback will lead to symptom reduction.

SUMMARY:
This is a prevention intervention study that will examine the efficacy of a smartphone-based intervention in decreasing cancer risk by targeting mental health risk factors of anxiety and depression.

DETAILED DESCRIPTION:
This prevention intervention study aims to examine the efficacy of a smartphone-based intervention in decreasing cancer risk by targeting mental health risk factors of anxiety and depression. The study will utilize a smartphone application called Mood Triggers, designed to provide personalized feedback on individuals' maintenance factors (i.e., "triggers") of their anxiety and depressive symptoms. Mood Triggers delivers ultra-brief interventions (less than 2 minutes long) where participants view videos introducing important skills to treat their anxiety and depression. The study targets middle-aged adults (40-64 years old) who meet current criteria for moderate to severe anxiety and/or depressive disorders. It will enroll an anticipated 100 participants in a single-group, open-label design, with the intervention lasting up to 12 weeks. The primary outcomes include changes in depression and anxiety symptoms, measured by the Patient Health Questionnaire-9 and the Generalized Anxiety Disorder-Q-IV Scale, respectively, as well as changes in cancer risk assessed by the World Cancer Research Fund/American Institute for Cancer Research Cancer Prevention Score.

ELIGIBILITY:
Inclusion Criteria:

1. Middle-aged adults (age 40 to 64).
2. fluent in English.
3. Able to provide informed consent.
4. Meets current criteria for an anxiety and/or depressive disorder with severity ranging from moderate to severe (based on the Patient Health Questionnaire - 9 and the Generalized Anxiety Disorder Questionnaire).
5. Owns a smartphone.

Exclusion Criteria:

1. Acute psychosis (based on the self-reported Structured Interview for Psychosis risk Syndromes, Prodromal Questionnaire - Brief version [SIPS PQ-B]).
2. Moderate to high suicidal ideation (based on a response of 2 or more on the PHQ-9 item-9).
3. History of bipolar disorder (based on the self-reported Mood Disorder Questionnaire [MDQ].
4. Past or current diagnoses of cancer.
5. Changes to treatments or medications in the past 30 days.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Changes in depression as assessed by Patient Health Questionnaire-9 | Baseline
  Possible PHQ-9 scores range from 0 to 27, with higher scores representing greater MDD symptom severity
Changes in depression as assessed by Patient Health Questionnaire-9 | 6 weeks post-baseline
  Possible PHQ-9 scores range from 0 to 27, with higher scores representing greater MDD symptom severity.
Changes in depression as assessed by Patient Health Questionnaire-9 | 12 weeks post-baseline
  Possible PHQ-9 scores range from 0 to 27, with higher scores representing greater MDD symptom severity
Change in anxiety symptoms as assessed by Generalized Anxiety Disorder- Q-IV Scale | At baseline
  Possible GAD-Q-IV scores range from 0 to 12, with higher scores representing greater GAD symptom severity
Change in anxiety symptoms as assessed by Generalized Anxiety Disorder- Q-IV Scale | 6 weeks post-baseline
  Possible GAD-Q-IV scores range from 0 to 12, with higher scores representing greater GAD symptom severity
Change in anxiety symptoms as assessed by Generalized Anxiety Disorder- Q-IV Scale | 12 weeks post-baseline
  Possible GAD-Q-IV scores range from 0 to 12, with higher scores representing greater GAD symptom severity
World Cancer Research Fund (WCRF)/ American Institute for Cancer Research (AICR) Cancer Prevention Score. | Up to 12 weeks after enrollment
  Minimum score: 0, Maximum score: 7-8 (8 for persons capable of breastfeeding). Greater scores suggest lower cancer risk.

SECONDARY OUTCOMES:
Smartphone estimates of sociability as mechanisms of change in cancer risk | Up to 12 weeks after enrollment
  Based on continuous passive mobile sensor data, sociability estimates will be based on the frequency of phone calls and texts.
Smartphone estimates of motion activity as mechanisms of change in cancer risk | Up to 12 weeks after enrollment
  Based on both activity levels based on the metabolic equivalent of task (MET) based on passively observed accelerometer data from the smartphone and daily movement based on geolocation data passively collected from the smartphone.
Diet as mechanism of change in cancer risk | Baseline, 6 weeks post-baseline, 12 weeks post-baseline
  Self-reported dietary intake will be recorded via entry of food intake in ASA24 and used when calculating WCRF/AICR cancer score. Diets rich in nutrients contribute to higher score (lower risk).
Momentary Assessment of Anxiety Symptom Changes | Up to 12 weeks after enrollment
  Thirteen items from a modified PHQ/GAD questionnaire will be used to measure daily anxiety and depression. Participants will rate answers on a 101 point scale ranging from 0-100 and is scaled from "Not at all" - "Constantly". Higher scores indicate generally more severe anxiety symptoms.
Momentary Assessment of Depression Symptom Changes | Up to 12 weeks after enrollment
  Thirteen items from a modified PHQ/GAD questionnaire will be used to measure daily anxiety and depression. Participants will rate answers on a 101 point scale ranging from 0-100 and is scaled from "Not at all" - "Constantly". Higher scores indicate generally more severe MDD symptoms.
Momentary Assessment of Behavioral Avoidance Symptom Changes | Up to 12 weeks after enrollment
  One item adapted from the Multidimensional Experiential Avoidance Questionnaire will be presented to measure daily changes in behavioral avoidance. A second item will be asked to measure self-reported changes in behavioral avoidance since the previous prompt.
Momentary Assessment of Hopelessness Symptom Changes | Up to 12 weeks after enrollment
  One item adapted from the Hopelessness Scale will be presented to gather a momentary measurement. A second momentary measurement will be presented to gather current self-report of feeling hopelessness.
Momentary Assessment of Arousal Symptom Changes | Up to 12 weeks after enrollment
  A self-report measure will ask current level of arousal on a sliding scale from "Sleepy" to "Active". Minimum or maximum values range from 0 (Sleepy) to 1 (Active).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Jacobson, PhD, Principal Investigator — Geisel School of Medicine, Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States